CLINICAL TRIAL: NCT03630978
Title: The Impact of Sarcopenia, Body Composition and Other Biometric Parameters on the Postoperative Outcomes of Patients Undergoing Liver Resection for Different Indications
Brief Title: Impact of Sarcopenia on Postoperative Outcomes of Patients Undergoing Liver Resection
Status: Completed | Type: Observational
Sponsor: San Camillo Hospital, Rome (Other)
Responsible Party: Principal Investigator, Giammauro Berardi, Resident in Surgery, Principal Investigator, San Camillo Hospital, Rome
Other Study IDs: 2018.01
Record Dates: First submitted 2018-08-11; First posted 2018-08-15 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Liver Neoplasms; Sarcopenia; Postoperative Complications
Keywords: hepatocellular carcinoma; colorectal liver metastases; non-colorectal liver metastases; focal nodular hyperplasia; liver hemangioma; liver cysts; surgical morbidity; surgical mortality; sarcopenia
MeSH Terms: conditions — Liver Neoplasms; Sarcopenia; Postoperative Complications; Carcinoma, Hepatocellular; Focal Nodular Hyperplasia | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver resection
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Major or minor, open or laparoscopic liver resection

SUMMARY:
The investigators will investigate the impact of different biometric parameters (Body mass index, sarcopenia, lean muscle mass, hand-grip strength, gait speed, fat composition) on the postoperative outcomes of patients undergoing liver resections.

Major and minor liver resections will be considered as well as open and minimally invasive techniques.

Benign and malignant indications will be included. Patients characteristics and perioperative variables will be considered for analysis.

Short-term outcomes will be evaluated focusing on 90-days morbidity and mortality and readmission rate.

DETAILED DESCRIPTION:
According to the null hypothesis, no difference in postoperative morbidity between the two groups would be expected. To calculate sample size, a 42% morbidity rate would be expected in sarcopenic patients while a 22% rate would be expected in the non-sarcopenic group. Considering a two-sided α=0.05 and β=0.1, the minimal sample size required to achieve statistical significance was 224 subjects. Considering a 10% drop-out rate of patients undergoing explorative laparoscopy or laparotomy without parenchymal resection a total of 249 patients will be required for completion of the study

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing open or laparoscopic liver resection
2. Patients undergoing major or minor liver resection
3. Patients undergoing liver resection for primary or secondary liver malignancies
4. Patients undergoing liver resections for benign diseases (cysts, adenoma, focal nodular hyperplasia, hemangioma) -

Exclusion Criteria:

1. Patients undergoing extrahepatic resection
2. Patients undergoing cyst fenestration or biopsies without liver resections
3. Patients with extrahepatic metastases
4. Patients undergoing explorative laparoscopy or laparotomy without parenchymal transection -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver resection for benign and malignant indications with CT scan imaging availability within 30 days before surgery.
  Of all the patients included in the study muscle function tests will be collected including handgrip strength, gait speed and fat composition.
  Preoperative antropometric, biochemical and disease presentation characteristics will be collected as well as operative details and postoperative outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Morbidity | within 90 days after surgery
  Patients experiencing medical or surgical complications after surgery

SECONDARY OUTCOMES:
Mortality | within 90 days after surgery
  Patients dying after surgery
Readmission rate | within 90 days after discharge
  patients readmitted to hospital after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Maria Ettorre, Prof, Study Director — San Camillo Hospital Spallanzani
Locations (1):
- San Camillo Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang G, Meng S, Li R, Ye J, Zhao L. Clinical significance of sarcopenia in the treatment of patients with primary hepatic malignancies, a systematic review and meta-analysis. Oncotarget. 2017 Jul 28;8(60):102474-102485. doi: 10.18632/oncotarget.19687. eCollection 2017 Nov 24. PMID 29254263
- [Result] Harimoto N, Yoshizumi T, Izumi T, Motomura T, Harada N, Itoh S, Ikegami T, Uchiyama H, Soejima Y, Nishie A, Kamishima T, Kusaba R, Shirabe K, Maehara Y. Clinical Outcomes of Living Liver Transplantation According to the Presence of Sarcopenia as Defined by Skeletal Muscle Mass, Hand Grip, and Gait Speed. Transplant Proc. 2017 Nov;49(9):2144-2152. doi: 10.1016/j.transproceed.2017.09.017. PMID 29149975
- [Result] Simonsen C, de Heer P, Bjerre ED, Suetta C, Hojman P, Pedersen BK, Svendsen LB, Christensen JF. Sarcopenia and Postoperative Complication Risk in Gastrointestinal Surgical Oncology: A Meta-analysis. Ann Surg. 2018 Jul;268(1):58-69. doi: 10.1097/SLA.0000000000002679. PMID 29373365